CLINICAL TRIAL: NCT03125720
Title: Image Fusion of SPECT MPI and Fluoroscopy Venography to Guide LV Lead Placement for Improved CRT Response (GUIDE-CRT II)
Acronym: GUIDE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Shanghai Zhongshan Hospital (Other); Shanghai Chest Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xijing Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); First People's Hospital of Hangzhou (Other); Anhui Provincial Hospital (Other Government); The Affiliated Hospital of Xuzhou Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); General Hospital of Shenyang Military Region (Other); Nanjing Medical University (Other); Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FirstNanjingMU001
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Heart Failure
Keywords: cardiac resynchronization therapy; chronic heart failure; image fusion-guided implantation; SPECT; venogram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUIDED group (Experimental): Image fusion of SPECT MPI and fluoroscopy venography to guide LV lead placement for improved CRT response in the guided group.
  Interventions: Other: Image fusion of SPECT MPI and fluoroscopy venography
- Control group (No Intervention): No Image fusion of SPECT MPI and fluoroscopy venography to guide LV lead placement for improved CRT response.

INTERVENTIONS:
Other: Image fusion of SPECT MPI and fluoroscopy venography — In this study, MPI-Fluoro Fusion tool is used to help the implanting physicians to precisely implant LV lead to the optimal/suboptimal venous segments in the guided group.
  Arms: GUIDED group

SUMMARY:
CRT response will be significantly better using image fusion of SPECT MPI and fluoroscopy venogram to guide LV lead placement at the latest activation segment without scar than standard-of-care implantation.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is final phase of a variety of cardiovascular diseases. Epidemiological data revealed that the morbidity of CHF is 0.9% in China, and there are 300,000 new CHF patients are diagnosed each year. Moreover, the total number of CHF patients exceeded 5.5 million throughout the country. Therefore, CHF has become a seriously social and public health problem in China.

Although medical treatment for CHF has achieved considerable progress, prognosis is still poor and mortality is high among end-stage HF patients. Since the 1990s, cardiac resynchronization therapy(CRT) has been applied to treat CHF, a large number of evidence-based medicine has shown that CRT brings great clinical effects; CRT mainly aims at delayed activation of left ventricular(LV) and stimulates LV in advance to restore the inter- and intra-ventricular synchrony. As a result, cardiac function, symptoms and quality of life in CHF patients improved, meanwhile mortality rate also decreases. At present, CRT is recommended in quite a number of CHF patients as class I indication. And yet, approximately 30%-40% of patients did not show response to CRT. Non-response to CRT has become a significant problem that must be solved. In recent years, researchers have tried LV multipoint pacing (MPP), transseptal left ventricular endocardial pacing and MitraClip to get some achievements. But these new techniques and CRT itself have two main failings:(1) Up to now, there is no specific suggestions about whether the patient's myocardium has too severe myocardial fibrosis and scar burden to be fit for CRT.(2)The LV mechanical dysynchronization will influence CRT effects. So far, screening CRT indications is primarily based on QRS morphology and duration on surface electrocardiogram.QRS duration≥120ms represents the presence of electrical dysynchronization, however, electrical dysynchronization is not equal to mechanical dysynchronization. The key point of CRT is to solve the mechanical dysynchronization, so estimating cardiac mechanical dysynchrony is important for predicting the CRT response; In addition, LV lead implantation site also exerts an effect on CRT response. The standard-of-care of LV lead implantation technique now just relays on coronary vein angiography showing the appropriate branch vein. This approach cannot guarantee LV lead is implanted in the latest activation site and the non-scar segment. Therefore, the following two issues are very important: how to evaluate the myocardiac scar and LV mechanical dyssynchronization using an objective, accurate, simple and economic method? and how to explore a new image which can guide LV lead to position at the latest activation and non-scar segment conveniently and accurately during procedure for improving CRT response rate? Myocardial perfusion image-phase analysis technique(MPI-PA) is a new non-invasive method to evaluate LV desynchronization,the latest activation site and myocardial scar burden. In recent years,Henneman MM and Adelstein EC reported PA technique detecting LV systolic desynchronization and LV scar burden influencing on CRT response respectively. Their study showed that the low CRT response is associated with the mild LV dyssynchrony and severe scar burden.The past five years,our center has completed a prospective, randomized, multi-center study of"SPECT guided LV Lead Placement for Incremental Benefits to CRT Efficacy"(GUIDE-CRT).We found that the CRT efficacy in SPECT-Guided group at 6 months after CRT implantation was better than that in standard-of-care implantation group(control group):the reduction in LVESV at 6 months in guided group is much more than that in control group(control 28.2ml vs guided group 48.2ml,P=0.029). The CRT response rate, defined as reduction in LVESV more than 15%, in guided group was 55.8% is higher than 47.8% in control group,but there was no statistic difference between two groups.The guiding mothodology of implanting LV lead in our previous study (GUIDE-CRT) was as following: implanter chose the branch vein to implant LV lead based on the recommended site by MPI-PA. Under this guidance, still much percentage of LV lead did not located in the recommended site. Therefore, in order to further improve the accuracy of SPECT guiding LV lead placement, our present study will use automatic fusion of coronary venogram with SPECT images to guide the implantation of LV lead precisely, and bringing incremental benefits to CRT efficacy.

This new study(GUIDE-CRT II) is a prospective, randomized, multi-center trial. Applying the new image fusion of SPECT MPI and coronary venogram to guide LV lead placement at the recommended optimal position, to achieve the precise localization, to avoid blindness of standard of care implantation methods and to improve response to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed informed consent
* moderate to severe HF (NYHA Class II, III or IV)
* LVEF ≤35%
* QRS duration ≥130 ms
* sinus rhythm

Exclusion Criteria:

* Patient is under a minimum age requirement (<18 years old)
* Patient has mechanical right heart valve
* Patient has experienced unstable angina, acute MI, CABG or PCI within the past 3 months
* Patient is on continuous or intermittent (i.e., more than two infusions per week) intravenous inotropic drug therapy
* Patient known to have chronic permanent atrial arrhythmias (i.e., cases of long-standing atrial fibrillation of greater than 1 year, including those in which cardioversion has not been indicated or attempted).
* Patient is enrolled in any other study
* Patient has a life expectancy of less than 12 months
* Women who are pregnant, or with child-bearing potential and who are not on a form of birth control
* Patient with CRT device implanted previously
* Patient has had a heart transplant
* Patient has third degree AVB with normal cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in LVESV | 6-month follow-up
  Changes in LVESV between baseline and 6-month follow-up (a continuous variable): LVESV will be assessed by echocardiography (Simpson's rule). Changes in LVESV will be compared between the two groups.

SECONDARY OUTCOMES:
CRT response rate | 6-month follow-up
  The proportion of the positive CRT response in each group. A positive CRT response is defined as reduction in LVESV by ≥15% and/or LVEF increase by ≥10% at 6-month follow-up as compared to the baseline.
Changes in LVEF | 6-month follow-up
  LVEF will be assessed by echocardiography (Simpson's rule) and compared between the baseline and 6-month follow-up. Changes in LVEF will be compared between the two groups.
Composite clinical response rate | 6-month follow-up
  A positive response is defined as decrease by ≥1 NYHA class and/or improvement in 6MWD by ≥10% and/or decrease in QOL score by ≥ 9 points at 6-month follow-up.
  * NYHA class: Changes in NYHA class at 6-month follow-up as compared to the baseline will be compared between the two groups.
  * 6MWD: Changes in 6MWD at 6-month follow-up as compared to the baseline will be compared between the two groups.
  * QOL: Changes in QOL score at 6-month follow-up as compared to the baseline will be compared between the two groups.
All-cause mortality and composite clinical endpoints | 6-month follow-up
  All-cause mortality,all-cause death and heart failure re-hospitalization by the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Zou, MD,Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (14):
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu Province People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital,Zhejiang University, Hangzhou, Zhejiang
  - First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Fu Wai Hospital, Beijing
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an
  - Xijing Hospital, Xi'an

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Result] Zhou W, Hou X, Piccinelli M, Tang X, Tang L, Cao K, Garcia EV, Zou J, Chen J. 3D fusion of LV venous anatomy on fluoroscopy venograms with epicardial surface on SPECT myocardial perfusion images for guiding CRT LV lead placement. JACC Cardiovasc Imaging. 2014 Dec;7(12):1239-48. doi: 10.1016/j.jcmg.2014.09.002. Epub 2014 Nov 5. PMID 25440593